CLINICAL TRIAL: NCT00678691
Title: An Eight Week, Double-Blind Efficacy Study of Armodafinil Augmentation to Alleviate Fibromyalgia Fatigue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Thomas L. Schwartz, M.D., Assoc Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ArmoFibro-001; NCT00568919 (obsolete NCT alias)
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia, Primary
Keywords: fibromyalgia; fatigue
MeSH Terms: conditions — Fibromyalgia; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A,1 (Experimental): armodafinil
  Interventions: Drug: armodafinil
- A,2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: armodafinil — 50-250mg/d
  Arms: A,1
Drug: placebo — matching placebo
  Arms: A,2

SUMMARY:
Armodafinil (NuvigilTM) is an isomer of a drug currently approved by the FDA for the treatment of fatigue secondary to narcolepsy, sleep apnea, and shift work sleep disorder called modafinil (ProvigilTM). There is considerable off label evidence for modafinil's ability to reduce fatigue related to multiple sclerosis, Parkinson's disease, cancer related fatigue, and depression related fatigue. There are preclinical studies showing that modafinil can alleviate fatigue secondary to medication side effects (diazepam, chlorpromazine). This multi-layered evidence base suggests that modafinil may be able to alleviate fatigue regardless of medical illness. Armodafinil now has four completed Phase III FDA regulatory studies revealing that it is well tolerated and effective for fatigue associated with obstructive sleep apnea (Effects of Armodafinil in the Treatment of Residual Excessive Sleepiness Associated with Obstructive Sleep Apnea/Hypopnea Syndrome: A 12-Week, Multicenter, Double-Blind, Randomized,Placebo-Controlled Study in nCPAP-Adherent Adults. Thomas Roth et al. Clinical Therapeutics/Volume 28, Number 5, 2006), shift work sleep disorder, and narcolepsy. Armodafinil is not yet FDA approved. It is felt to be a cleaner, safer, more potent isomer. Theoretically, fatigue is interpreted and possibly dictated centrally and armodafinil's proposed mechanism (similar to that of modafinil) of elevating central histamine activity may allow the brain to interpret a lower fatigue state, thus allowing patients to function better during the day with less peripheral fatigue.

Fibromyalgia (FM) is an illness that may involve medical, rheumatological, autoimmune, sleep, endocrine and psychiatric pathology. It is a syndrome of recurrent pain at trigger points. Greater than 90% of these patients will report fatigue as a key symptom as well. There are several investigation lines into the treatment of FM induced pain. Exercise, behavioral therapy, amitryptiline, duloxetine, tramadol, sodium oxybate all have randomized trials and almost all focus on pain. There are very few studies, if any, that look at FM induced fatigue which certainly ads to FM patients' daily incapacity and lowered productivity/quality of life.

Armodafinil is a drug with minimal adverse effects (headache, insomnia, GI distress, anxiety, dry mouth, dizziness and an assumed low level addiction which is comparable to modafinil) which is well tolerated in current regulatory studies. It may have a safer tolerability profile than the FM medications noted above. As modafinil is often studied and often added as an augmentation agent to patients' regimens who suffer from fatigue in other medical illnesses, the authors feel that armodafinil would also be effective in this population. The authors wish to conduct a study to determine if armodafinil is safe and tolerable in the treatment of FM induced fatigue. This initial controlled study may allow for continued regulatory studies with this product in FM subjects. We propose a double-blind placebo controlled study to determine if armodafinil is safe and effective in reversing FM induced fatigue.

ELIGIBILITY:
Inclusion Criteria:

* If possible, 60 subjects will be included in this study.
* All males/females of any race are eligible if aged between 18 and 65 and
* Subjects must speak English and have capacity to receive and utilize informed consent
* Agree to use barrier method contraception or are infertile x2 years due to medical condition or surgery
* Have been formally diagnosed by a Board Certified Rheumatologist using the ACR 1990 research criteria for fibromylagia
* Report that fatigue, in addition to FM pain is a key distressing symptom of their FM
* Have a score of >4 on the Brief Fatigue Inventory (BFI)
* Women of child bearing potential must agree to use barrier contraception as armodafinil may decrease the effectiveness of oral contraceptives

Exclusion Criteria:

* Exclusion: Subjects cannot
* Be pregnant or be attempting to conceive at present (urine bHCG must be negative)
* Have an active substance abuse problem with last use within the past 180 days (outside of nicotine)
* Use other stimulating medication ie stimulants, caffeine products (this refers to OTC stimulants OR patients clinically tolerant to and withdrawing from caffeinated beverages, bupropion, desipramine, etc UNLESS said drug has been in steady dosing for >4 weeks
* Have a known medical condition outside of FM that causes fatigue (i.e. obstructive apnea, hypothyroidism, depression, etc)
* Have a known medical condition or other medication use that relatively contraindicates armodafinil use (ie substance abuse, sensitivity to armodafinil, known cardiac abnormalities of left ventricular hypertrophy, recent MI, mitral valve prolapse dependent on stimulant use, history of psychosis
* Has a prior history of modafinil use and failure
* Be receiving daytime sedating medication with clear chronological impact on fatigue UNLESS fatigue predates sedating medication or said medication has been steadily dosed > 4 weeks
* Medications that induce/inhibit p450 3A4 as they may alter armodafinil plasma levels, and vica versa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were easily recruited and screened for study entry
Pre-assignment Details: Subjects were exluded after informed consent if medical confounding variables or safety variables were found
Groups:
- A,1 Armodafinil Study Drug 50-250mg Flexible Dose: armodafinil
- A,2 Matching Placebo: placebo
Period: Overall Study
Arm/Group | A,1 Armodafinil Study Drug 50-250mg Flexible Dose | A,2 Matching Placebo
Started | 27 | 28
Completed | 21 | 24
Not Completed | 6 | 4
Not completed — Adverse Event | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- A,1 Armodafinil Study Drug: armodafinil
- Total: Total of all reporting groups
Arm/Group | A,1 Armodafinil Study Drug | A,2 Matching Placebo | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (4) | 47 (4) | 49 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Brief Fatigue Inventory
Description: This scale measures overall fatigue due to medical illness. range is 0-80 with 80 being severe fatigue
Time Frame: 8 weeks
Population: last observation carried forward after power analysis calculated
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A,1 Armodafinil Study Drug | A,2 Matching Placebo
Number analyzed (Participants) | 27 | 28
units on a scale | 2.86 (.149) | 4.29 (.144)
Statistical Analysis 1: Comparison: A,1 Armodafinil Study Drug vs A,2 Matching Placebo; Authors expected armodafinal to work better than placebo reducing BFI scale scores by 30%. A piecewise statistical model was used to compare baseline scores against those over through week 8. Piecewise results for between group differences for BFI Scores: P=.390 (baseline through week 5), p=.775 (week 5 - week 8); Test type: Superiority or Other; p < 0.05, piecewise model — all p-values come from one model analysis and are therefore included in free text as such; A piecewise statistical model results for between group differences: P=.390 (baseline through week 5), p=.775 (week 5 - week 8

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | A,1 Armodafinil Study Drug | A,2 Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 9/27 | 8/28
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | A,1 Armodafinil Study Drug (N=27) | A,2 Matching Placebo (N=28)
headache (Vascular disorders) | 4 | 3
dry mouth (Gastrointestinal disorders) | 3 | 3
Poor Concentration (Psychiatric disorders) | 2 | 2/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No